CLINICAL TRIAL: NCT04939428
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of MK-4482 for the Prevention of COVID-19 (Laboratory-confirmed SARS-CoV-2 Infection With Symptoms) in Adults Residing With a Person With COVID-19
Brief Title: Study of MK-4482 for Prevention of Coronavirus Disease 2019 (COVID-19) in Adults (MK-4482-013)
Acronym: MOVe-AHEAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4482-013; MK-4482-013 (Other: MSD); jRCT2031210281 (Registry Identifier: jRCT (Japan Registry of Clinical Trials)); PHRR211007-003980 (Registry Identifier: PHRR); 2021-000904-39 (EudraCT Number)
Record Dates: First submitted 2021-06-24; First posted 2021-06-25 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Molnupiravir (Experimental): Participants take molnupiravir 800 mg every 12 hours (Q12H) on Days 1 to 5.
  Interventions: Drug: Molnupiravir
- Placebo (Placebo Comparator): Participants take placebo Q12H on Days 1 to 5.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Molnupiravir — Four molnupiravir 200 mg capsules taken by mouth.
  Other Names: MK-4482
  Arms: Molnupiravir
Drug: Placebo — Placebo capsule matched to molnupiravir 200 mg capsules taken by mouth.
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess if the study medication (molnupiravir, MK-4482) will prevent symptomatic coronavirus disease 2019 (COVID-19) in adults who live with someone with confirmed COVID-19 infection. This is a phase 3, multicenter, randomized, double-blind, placebo-controlled study; half of the study participants will receive molnupiravir twice daily by mouth and the other half will receive a placebo. The primary objectives of the study are to determine if molnupiravir prevents symptomatic COVID-19 disease and to evaluate its safety and tolerability. All participants who develop COVID-19 during the study are still eligible for any COVID-19 treatment recommended by their doctor.

ELIGIBILITY:
Inclusion Criteria:

* Lives in a household with an index case where the index case is a person with documented COVID-19 (laboratory-confirmed SARS-CoV-2 infection with symptoms case) and must have 1) a first detectable SARS-CoV-2 test result from a sample collected within ≤5 days prior to randomization of the participant, and 2) at least 1 symptom attributable to COVID-19 (e.g., fever, difficulty breathing)
* Does not have confirmed or suspected COVID-19
* Is willing and able to take oral medication
* For males, agrees to be abstinent from penile-vaginal intercourse OR agrees to use a highly effective contraceptive method while receiving study drug and for ≥3 months after the last dose of study drug
* Is female and not pregnant/breastfeeding and at least one of the following applies during the study and for ≥4 days after: is not a woman of childbearing potential (WOCBP), is a WOCBP and uses highly effective contraception (low user dependency method OR a user dependent hormonal method in combination with a barrier method), or is a WOCBP who is abstinent from heterosexual intercourse

Exclusion Criteria:

* Has a prior history of laboratory-confirmed SARS-CoV-2 infection (with or without symptoms) within 6 months prior to randomization
* Has either of the following: human immunodeficiency virus (HIV) with a recent viral load >50 copies/mL (regardless of CD4 count) or an acquired immunodeficiency syndrome (AIDS)-defining illness
* Has a history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection with any of the following: cirrhosis, end-stage liver disease, hepatocellular carcinoma; aspartate transaminase (AST) and/or (ALT) >3x upper limit of normal at screening
* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator
* Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments including but not limited to participants with conditions that could limit gastrointestinal absorption of capsule contents
* Has received, is taking, or is anticipated to require any prohibited therapies
* Has received a COVID-19 vaccination with the first dose ≥7 days prior to randomization
* Is unwilling to abstain from participating in another interventional clinical study through Day 29 with an investigational compound or device, including those for COVID-19 therapeutics
* Is living in a household with >10 people

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2441 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (226):
- United States (59):
  - Cahaba Research, Inc. ( Site 2523), Birmingham, Alabama
  - The Institute for Liver Health DBA Arizona Clinical Trials ( Site 2484), Mesa, Arizona
  - The Institute for Liver Health DBA Arizona Clinical Trials ( Site 2448), Tucson, Arizona
  - Hope Clinical Research ( Site 2400), Canoga Park, California
  - Carbon Health ( Site 2515), Carlsbad, California
  - UCSF Fresno ( Site 2528), Fresno, California
  - ASCADA Research, LLC ( Site 2516), Fullerton, California
  - Marvel Clinical Research ( Site 2490), Huntington Beach, California
  - National Research Institute ( Site 2452), Los Angeles, California
  - Valley Clinical Trials Inc. ( Site 2406), Northridge, California
  - Carbon Health ( Site 2514), Oakland, California
  - University of California Davis ( Site 2497), Sacramento, California
  - Millennium Clinical Trials ( Site 2468), Simi Valley, California
  - Future Innovative Treatments, LLC ( Site 2471), Colorado Springs, Colorado
  - Emerson Clinical Research Institute ( Site 2457), Washington D.C., District of Columbia
  - Synergy Healthcare ( Site 2521), Bradenton, Florida
  - Accel Research Sites-DeLand Clinical Research Unit ( Site 2535), DeLand, Florida
  - Velocity Clinical Research, Hallandale Beach ( Site 2485), Hallandale, Florida
  - Indago Research and Health Center Inc ( Site 2412), Hialeah, Florida
  - Advanced Research For Health Improvement LLC ( Site 2436), Immokalee, Florida
  - Clinical Site Partners, LLC d/b/a CSP Miami ( Site 2508), Miami, Florida
  - CDC Research Institute, LLC ( Site 2540), Port Saint Lucie, Florida
  - Clinical Research Trials of Florida ( Site 2402), Tampa, Florida
  - Clinical Site Partners, LLC d/b/a CSP Miami ( Site 2425), Winter Park, Florida
  - Balanced Life Healthcare Solutions/SKYCRNG ( Site 2539), Lawrenceville, Georgia
  - Chicago Clinical Research Institute Inc ( Site 2454), Chicago, Illinois
  - Rush University Medical Center ( Site 2510), Chicago, Illinois
  - Southern Clinical Research Associates ( Site 2542), Metairie, Louisiana
  - MedPharmics, LLC ( Site 2443), Metairie, Louisiana
  - Institute of Human Virology ( Site 2504), Baltimore, Maryland
  - Centennial Medical Group ( Site 2435), Elkridge, Maryland
  - Jadestone Clinical Research, LLC ( Site 2530), Silver Spring, Maryland
  - Michigan Center of Medical Research ( Site 2445), Farmington Hills, Michigan
  - Michigan Center of Medical Research ( Site 2525), Lathrup Village, Michigan
  - Allina Health Infectious Diseases Research Clinic ( Site 2507), Minneapolis, Minnesota
  - Prime Health and Wellness/SKYCRNG ( Site 2538), Fayette, Mississippi
  - Quinn Healthcare/Skycrng ( Site 2537), Ridgeland, Mississippi
  - University of Missouri Hospital ( Site 2486), Columbia, Missouri
  - Mercury Street Medical Group PLLC ( Site 2476), Butte, Montana
  - University of Nebraska Medical Center ( Site 2430), Omaha, Nebraska
  - Excel Clinical Research, LLC ( Site 2404), Las Vegas, Nevada
  - ID Care ( Site 2466), Hillsborough, New Jersey
  - Amici Clinical Research LLC ( Site 2426), Raritan, New Jersey
  - AXCES Research Group ( Site 2437), Santa Fe, New Mexico
  - Montefiore Medical Center ( Site 2503), The Bronx, New York
  - ECU Adult Specialty Care ( Site 2415), Greenville, North Carolina
  - The Lindner Center for Research and Education at The Christ Hospital ( Site 2517), Cincinnati, Ohio
  - Dayton Clinical Research ( Site 2488), Dayton, Ohio
  - Cherokee Nation WW Hastings Indian Hospital/Cherokee Nation Health Services ( Site 2459), Tahlequah, Oklahoma
  - Preferred Clinical Research ( Site 2470), Pittsburgh, Pennsylvania
  - Velocity Clinical Research-Providence ( Site 2432), East Greenwich, Rhode Island
  - Tribe Clinical Research, LLC ( Site 2409), Greenville, South Carolina
  - PharmaTex Research, LLC ( Site 2541), Amarillo, Texas
  - TTS Research ( Site 2433), Boerne, Texas
  - Houston Methodist Hospital ( Site 2463), Houston, Texas
  - Santa Clara Family Clinic ( Site 2462), Houston, Texas
  - Crossroads Clinical Research LLC ( Site 2451), Victoria, Texas
  - TPMG Clinical Research ( Site 2495), Williamsburg, Virginia
  - Covid-19 Clinical Research Center (CCRC) ( Site 2421), Seattle, Washington
- Argentina (8):
  - Sanatorio de la Trinidad Mitre ( Site 0108), CABA, Buenos Aires
  - Mautalen Salud e Investigacion ( Site 0103), Caba, Buenos Aires
  - Hospital Italiano de Buenos Aires ( Site 0102), CABA, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0105), Mar del Plata, Buenos Aires
  - Clinica Independencia ( Site 0104), Munro, Buenos Aires
  - Grupo Oroño Centro medico San Nicolas ( Site 0109), San Nicolás de los Arroyos, Buenos Aires
  - Instituto Medico de la Fundacion Estudios Clinicos ( Site 0106), Rosario, Santa Fe Province
  - CEMIC ( Site 0101), Buenos Aires
- Brazil (7):
  - Fundaçao de Medicina Tropical Doutor Heitor Vieira Dourado ( Site 0303), Manaus, Amazonas
  - Faculdade de Medicina da Universidade Federal de Mato Grosso do Sul - UFMS ( Site 0305), Campo Grande, Mato Grosso do Sul
  - Hospital Nossa Senhora das Gracas ( Site 0310), Curitiba, Paraná
  - Oncosite-Centro de Pesquisa Clinica em Oncologia ( Site 0300), Ijuí, Rio Grande do Sul
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 0312), São José do Rio Preto, São Paulo
  - Centro de Referencia Professor Helio Fraga - FIOCRUZ/RJ ( Site 0314), Rio de Janeiro
  - Centro de Referência e Treinamento DST/AIDS ( Site 0301), São Paulo
- Bulgaria (3):
  - Medical Center Hera EOOD ( Site 3001), Sofia, Sofia (stolitsa)
  - Medical Center Hera Kyustendi EOOD ( Site 3003), Kyustendil
  - Medical Center Hera EOOD - Montana branch ( Site 3002), Montana
- Colombia (10):
  - Fundacion Centro de Investigacion Clinica CIC ( Site 0402), Medellín, Antioquia
  - Centro Cientifico Asistencial Jose Luis Accini ( Site 0412), Barranquilla, Atlántico
  - Clinica de la Costa Ltda. ( Site 0407), Barranquilla, Atlántico
  - Caja de Compensacion Familiar CAFAM ( Site 0403), Bogotá, Bogota D.C.
  - Hospital Universitario Clinica San Rafael ( Site 0410), Bogota, Cundinamarca
  - Healthy Medical Center S.A.S ( Site 0413), Zipaquirá, Cundinamarca
  - Oncomedica S.A. ( Site 0406), Montería, Departamento de Córdoba
  - Fundacion Centro de Investigaciones Clinicas CARDIOMET ( Site 0409), Pereira, Risaralda Department
  - Instituto Neumologico del Oriente S.A. ( Site 0408), Bucaramanga, Santander Department
  - Fundacion Valle del Lili ( Site 0405), Cali, Valle del Cauca Department
- Unidad de Aislamiento del Centro de Obstetricia y Ginecologia ( Site 2650), Santo Domingo, Nacional, Dominican Republic
- Egypt (6):
  - Masri - CRC - Ain Shams University ( Site 2900), Cairo, Cairo Governorate
  - Masri - CRC - Ain Shams University ( Site 2910), Cairo, Cairo Governorate
  - National Hepatology and Tropical Medicine Research Institute ( Site 2930), Cairo, Cairo Governorate
  - Air Force Specialized Hospital Clinical Research Center ( Site 2920), Cairo, Cairo Governorate
  - National Center for allergies and chest ( Site 2940), Giza, Giza Governorate
  - Imbaba Fevers Hospital ( Site 2945), Giza, Giza Governorate
- France (5):
  - Maison de Sante Universitaire La Providence ( Site 0506), Toulouse, Haute-Garonne
  - CHU de la Reunion - Groupe Hospitalier Sud ( Site 0508), Saint-Pierre, La Reunion
  - CHU Martinique ( Site 0511), Fort-de-France, Martinique
  - Maison de santé du Pays Neufchatelois ( Site 0507), Neufchâtel-en-Bray, Seine-Maritime
  - Hôpital Pitié - Salpêtrière ( Site 0501), Paris, Île-de-France Region
- Guatemala (5):
  - Centro de Investigaciones Pediatricas ( Site 0703), Guatemala City
  - Unidad de Diagnostico Cardiologico ( Site 0701), Guatemala City
  - Clínica Médica Especializada en Pediatría e Infectología Pediátrica - Dr. Mario Melgar ( Site 0702), Guatemala City
  - Clinica Privada ( Site 0705), Guatemala City
  - Private Clinic - Dr. Hugo Pezzarossi ( Site 0704), Guatemala City
- Hungary (8):
  - LONA MEDIC Kft ( Site 0804), Orosháza, Bekes County
  - Debreceni Egyetem Klinikai Kozpont- Infektologiai Klinika ( Site 0824), Debrecen, Hajdú-Bihar
  - Bugat Pal Korhaz ( Site 0817), Gyöngyös, Heves County
  - Medifarma-98 Kft. ( Site 0808), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - DRC Gyogyszervizsgalo Kozpont Kft. ( Site 0801), Balatonfüred, Veszprém megye
  - Obudai Egeszsegugyi Centrum - OEC ( Site 0821), Budapest
  - Strazsahegy Medicina Bt ( Site 0823), Budapest
  - Obudai Egeszsegugyi Centrum - Zalaegerszeg ( Site 0819), Zalaegerszeg
- Japan (8):
  - IUHW Narita Hospital ( Site 1105), Narita, Chiba
  - National Hospital Organization Okinawa National Hospital ( Site 1109), Ginowan, Okinawa
  - Social Medical Corporation Yuuaikai Yuuai Medical Center ( Site 1108), Tomigusuku, Okinawa
  - Chiba Aoba Municipal Hospital ( Site 1100), Chiba
  - Global Healthcare Clinic ( Site 1106), Tokyo
  - Den-en-chofu family clinic ( Site 1104), Tokyo
  - Center Hospital of the National Center for Global Health and Medicine ( Site 1101), Tokyo
  - Sekino Hospital ( Site 1110), Tokyo
- Kenya (3):
  - Center for Clinical Research (CCR) KEMRI ( Site 1929), Nairobi, Nairobi City
  - Partners in Health Research and Development PHRD ( Site 1928), Nairobi, Nairobi City
  - KEMRI-CMR-RCTP- Kenya Medical Research Institute Kisumu ( Site 1925), Kisumu
- Malaysia (2):
  - Hospital Raja Perempuan Zainab II ( Site 2851), Kota Bharu, Kelantan
  - Klinik Kesihatan Masjid Tanah ( Site 2850), Masjid Tanah, Melaka
- Mexico (13):
  - Morales Vargas Centro de Investigacion, S.C. ( Site 1318), León, Guanajuato
  - Hospital General de Acapulco ( Site 1319), Acapulco de Juárez, Guerrero
  - Instituto Jalisciense de Metabolismo SC ( Site 1314), Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 1308), Mexico City, Mexico City
  - Centro Médico Universitario ( Site 1316), Cuernavaca, Morelos
  - CHRISTUS - LATAM HUB CENTER OF EXCELLENCE AND INNOVATION S.C. ( Site 1315), General Escobedo, Nuevo León
  - Centro de Investigacion y Avances Medicos Especializados -CIAME ( Site 1301), Cancún, Quintana Roo
  - Köhler & Milstein Research S.A. de C.V. ( Site 1300), Mérida, Yucatán
  - Centro de Investigacion Medica Aguascalientes ( Site 1305), Aguascalientes
  - ICARO Investigaciones en Medicina ( Site 1313), Chihuahua City
  - Medica Sur S.A.B de C.V. ( Site 1303), Mexico City
  - Oaxaca Site Management Organization S.C. ( Site 1304), Oaxaca City
  - Arké SMO S.A de C.V ( Site 1306), Veracruz
- Peru (7):
  - Policlínico Especializado en Neurología - Unid. Inv. Neurológica ( Site 1403), La Perla, Qallaw
  - Clínica Ricardo Palma ( Site 1406), Lima
  - Asociacion Civil por la Salud ( Site 1411), Lima
  - Investigaciones Medicas en Salud - INMENSA ( Site 1401), Lima
  - Asociacion Civil IMPACTA Salud y Educacion - Sede San Miguel ( Site 1410), Lima
  - Clinica Providencia ( Site 1400), Lima
  - Instituto de Investigacion Nutricional - Anexo Huascar ( Site 1404), Lima
- Philippines (3):
  - Asian Hospital and Medical Center ( Site 1503), Muntinlupa, National Capital Region
  - Quirino Memorial Medical Center ( Site 1501), Quezon City, National Capital Region
  - Health Index Multi-Specialty and Lying -in Clinic ( Site 1504), Cavite
- Romania (8):
  - Centrul Medical Unirea SRL ( Site 1707), Cluj-Napoca, Cluj
  - S.C Materna Care SRL ( Site 1702), Timișoara, Timiș County
  - Centrul Medical Unirea ( Site 1705), Brasov
  - Centrul Medical Unirea SRL Bucuresti ( Site 1706), Bucharest
  - Delta Heath Care S.R.L ( Site 1708), Bucharest
  - SC Policlinica CCBR SRL. Bucuresti ( Site 1704), Bucharest
  - Centrul Medical Unirea SRL Constanta ( Site 1703), Constanța
  - Centrul Medical Unirea SRL IASI ( Site 1701), Iași
- Russia (16):
  - FSBI Central Hospital with Policlinics ( Site 1807), Moscow, Moscow
  - Infectious Clinical Hospital # 1 ( Site 1834), Moscow, Moscow
  - SPb SBHI. City outpatient clinic No.44 ( Site 1830), Saint Petersburg, Sankt-Peterburg
  - SPb SBHI City outpatient clinic 112 ( Site 1829), Saint Petersburg, Sankt-Peterburg
  - Medical Research Institute LLC. ( Site 1814), Saint Petersburg, Sankt-Peterburg
  - Limited liability company "Scientific research center Eco-safety" ( Site 1809), Saint Petersburg, Sankt-Peterburg
  - Smorodintsev Research Institute of Influenza ( Site 1833), Saint Petersburg, Sankt-Peterburg
  - City Polyclinic #88 ( Site 1808), Saint Petersburg, Sankt-Peterburg
  - Nikolaevskaya hospital ( Site 1810), Saint Petersburg, Sankt-Peterburg
  - SPb SBHI City outpatient clinic 4 ( Site 1831), Saint Petersburg, Sankt-Peterburg
  - LLC -Medical Center . Capital-Polis ( Site 1825), Saint-Petrsburg, Sankt-Peterburg
  - St.Petersburg Outpatient Clinic No. 109 ( Site 1818), Saint-Petrsburg, Sankt-Peterburg
  - Smolensk State Medical Academy ( Site 1803), Smolensk, Smolensk Oblast
  - Republican Clinical Infectious Hospital n.a. A.F. Agafonov ( Site 1802), Kazan', Tatarstan, Respublika
  - Voronezh Regional Clinical Hospital #1 ( Site 1823), Voronezh, Voronezskaja Oblast
  - LLC -Clinic of modern medicine of Doctor Bogorodskaya ( Site 1828), Yaroslavl, Yaroslavl Oblast
- South Africa (18):
  - IATROS International ( Site 1921), Bloemfontein, Free State
  - REIMED Reiger Park ( Site 1910), Boksburg, Gauteng
  - Midrand Medical Centre ( Site 1913), Halfway House, Gauteng
  - Wits Health Consortium. Clinical HIV Research Unit ( Site 1923), Johannesburg, Gauteng
  - Right To Care Research - Esizayo ( Site 1907), Johannesburg, Gauteng
  - DJW Navorsing ( Site 1915), Krugersdorp, Gauteng
  - Zinakekele Medical Centre ( Site 1926), Moloto, Gauteng
  - Mzansi Ethical Research Centre ( Site 1918), Mpumalanga, Gauteng
  - Global Clinical Trial Centre ( Site 1904), Pretoria, Gauteng
  - Jongaie Research ( Site 1900), Pretoria West, Gauteng
  - Dr Jugnundun & Partners ( Site 1905), Durban, KwaZulu-Natal
  - Enhancing Care Foundation-DICRS ( Site 1922), Durban, KwaZulu-Natal
  - Private Practice - Dr. Neyaseelan Gounden ( Site 1911), Durban, KwaZulu-Natal
  - Limpopo Clinical Research Initiative ( Site 1901), Thabazimbi, Limpopo
  - TASK Applied Science ( Site 1920), Cape Town, Western Cape
  - DTHF Masiphumelele Clinical Research Site ( Site 1919), Cape Town, Western Cape
  - Be Part Yoluntu Centre ( Site 1914), Paarl, Western Cape
  - Paarl Research Centre ( Site 1924), Paarl, Western Cape
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol ( Site 2010), Badalona, Barcelona
  - CAP Centelles ( Site 2011), Centelles, Barcelona
  - Hospital de Alcorcon ( Site 2003), Alcorcón, Madrid, Comunidad de
  - C.S. Vallcarca-Sant Gervasi ( Site 2000), Barcelona
  - CAP de Sardenya ( Site 2009), Barcelona
  - Hospital Universitario Infanta Leonor ( Site 2002), Madrid
  - Hospital Universitario La Paz ( Site 2024), Madrid
- Thailand (5):
  - HIV-NAT AIDS Research Centre ( Site 2804), Bangkok, Bangkok
  - Chulabhorn Hospital ( Site 2801), Lak Si, Bangkok
  - Rajavithi Hospital ( Site 2803), Ratchathewi, Bangkok
  - The Golden Jubilee Medical Center ( Site 2800), Phutthamonthon, Changwat Nakhon Pathom
  - Songklanagarind Hospital ( Site 2802), Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (11):
  - Atakent Acibadem Hastanesi ( Site 2103), Halkali/K.cekmece, Istanbul
  - Ankara Universitesi Ibni Sina Hastanesi ( Site 2101), Ankara
  - Hacettepe Universitesi Tip Fakultesi ( Site 2102), Ankara
  - Gazi Universitesi Tip Fakultesi Hastanesi ( Site 2106), Ankara
  - Ankara Sehir Hastanesi ( Site 2111), Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi ( Site 2110), Istanbul
  - Medipol Universite Hastanesi ( Site 2108), Istanbul
  - Basaksehir Cam ve Sakura City Hospital ( Site 2112), Istanbul
  - Sancaktepe Prof Dr Ilhan Varank EAH-Prof Dr Feriha Oz Hastanesi ( Site 2113), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 2105), Izmir
  - Sakarya Universitesi Egitim ve Arastirma Hastanesi ( Site 2107), Sakarya
- Ukraine (13):
  - Ivano-Frankivsk Regional Clinical Infectious Diseases Hospital ( Site 2232), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Regional Phthisiopulmonological Center ( Site 2203), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - NPME -Central Clinical Hospital of Ivano-Frankivsk City Council ( Site 2204), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Non profit municipal enterprise City hospital student of Kharkiv city council ( Site 2229), Kharkiv, Kharkivs’ka Oblast’
  - PCNE Kharkiv City polyclinic 9 of the Kharkiv City Council ( Site 2201), Kharkiv, Kharkivs’ka Oblast’
  - Limited Liability Company Medical center Healthy Happy ( Site 2225), Kyiv, Kyivska Oblast
  - MNPE Consultative-Diagnostic Centre of Desnyanskyi District of Kyiv ( Site 2205), Kyiv, Kyivska Oblast
  - Kyiv railway clinical hospital 2 of Branch Health center ( Site 2207), Kyiv, Kyivska Oblast
  - Municipal Noncommercial Enterprise Lviv 4th City Clinical Hospital ( Site 2200), Lviv, Lviv Oblast
  - Odesa Regional Center of Socially Significant Diseases ( Site 2230), Odesa, Odesa Oblast
  - MNCE -Odesa regional clinical hospital of Odesa regional council ( Site 2226), Odesa, Odesa Oblast
  - Municipal Enterprise Poltava Regional Clinical Infectious Hospital ( Site 2227), Poltava, Poltava Oblast
  - Medical Clinical Investigational Center of Medical Center Health Clinic ( Site 2210), Vinnytsia, Vinnytsia Oblast

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Alpizar SA, Accini J, Anderson DC, Eysa B, Medina-Pinon I, Ohmagari N, Ostrovskyy MM, Aggrey-Amable A, Beck K, Byrne D, Grayson S, Hwang PMT, Lonchar JD, Strizki J, Xu Y, Paschke A, De Anda CS, Sears PS; MOVe-AHEAD study group. Molnupiravir for intra-household prevention of COVID-19: The MOVe-AHEAD randomized, placebo-controlled trial. J Infect. 2023 Nov;87(5):392-402. doi: 10.1016/j.jinf.2023.08.016. Epub 2023 Sep 9. PMID 37690669
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26072&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only eligible participants without confirmed or suspected coronavirus disease 2019 (COVID-19) were enrolled within a 5-day period of the index case's first positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test result and COVID-19 symptoms onset.
Pre-assignment Details: Index cases were enrolled but did not receive study treatment upon randomization and with the exception of characteristics collected at baseline and optional exploratory swab collection, no other data were collected.Index participants were not followed up for survival and no mortality data were collected per protocol.Index cases were not included in protocol specified outcome measure data collection.
Groups:
- Molnupiravir: Participants were treated with molnupiravir 800 mg every 12 hours (Q12H) on Days 1 to 5.
- Placebo: Participants were given placebo Q12H on Days 1 to 5.
- Index Participants: Index case was a participant with documented COVID-19 infection. Index participants were enrolled but did not receive study intervention. Index participants resided in the same household as enrolled participants who received study intervention.
Period: Overall Study
Arm/Group | Molnupiravir | Placebo | Index Participants
Started | 768 | 771 | 902
Treated | 763 | 765 | 0
Completed | 750 | 751 | 0
Not Completed | 18 | 20 | 902
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 5 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Randomized By Mistake Without Study Treatment | 1 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 11 | 0
Not completed — Unkown | 6 | 3 | 0
Not completed — Discotinued per protocol | 0 | 0 | 902

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Molnupiravir | Placebo | Index Participants | Total
Number analyzed (Participants) | 768 | 771 | 902 | 2441
Age, Continuous [Median (Standard Deviation); unit: years] | 37.0 (15.6) | 37.0 (15.5) | 38.0 (17.7) | 37.0 (15.6)
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 76 | 76
  Adults (18-49 years) | 563 | 568 | 548 | 1679
  From 50 to 64 years | 144 | 141 | 199 | 484
  From 65 to 74 years | 35 | 44 | 54 | 133
  >=75 years | 26 | 18 | 25 | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 366 | 342 | 541 | 1249
  Male | 402 | 429 | 361 | 1192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 323 | 340 | 341 | 1004
  Not Hispanic or Latino | 445 | 430 | 552 | 1427
  Unknown or Not Reported | 0 | 1 | 9 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 85 | 90 | 80 | 255
  Asian | 48 | 40 | 62 | 150
  Native Hawaiian or Other Pacific Islander | 1 | 4 | 2 | 7
  Black or African American | 62 | 60 | 77 | 199
  White | 453 | 446 | 552 | 1451
  More than one race | 119 | 129 | 128 | 376
  Unknown or Not Reported | 0 | 2 | 1 | 3
Stratification Factor at Randomization Collected via IRT: Household Size [Count of Participants; unit: Participants] — Population: Per protocol study specific charachteristics data was not collected for index cases as no study specific assessments were done.
  Participants
    number analyzed (Participants) | 768 | 771 | 0 | 1539
    <=3 | 269 | 271 | 0 | 540
    >=3 | 499 | 500 | 0 | 999
Stratification Factor at Randomization Collected via IRT: Age Group [Count of Participants; unit: Participants] — Population: Per protocol study specific charachteristics data was not collected for index cases as no study specific assessments were done.
  Participants
    number analyzed (Participants) | 768 | 771 | 0 | 1539
    <=60 | 680 | 680 | 0 | 1360
    >=60 | 88 | 91 | 0 | 179

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Undetectable SARS-CoV-2 in Baseline Nasopharyngeal (NP) Swabs and Developed COVID-19 (Laboratory-Confirmed SARS-CoV-2 Infection With Symptoms) Through Day 14
Description: Percentage of participants who had undetectable SARS-CoV-2 in baseline NP swabs and developed COVID-19 (laboratory-confirmed SARS-CoV-2 infection with symptoms) through Day 14 were reported.
Time Frame: Day 14
Population: Efficacy analysis was conducted on the mITT (modified intent to treat) population consisting of all randomized participants who received at least 1 dose of study intervention. Index participants were not included in OM analysis per protocol.
Measure: Number; unit: Percentage of Participants
Arm/Group | Molnupiravir | Placebo
Number analyzed (Participants) | 630 | 634
Percentage of Participants | 41 | 54
Statistical Analysis 1: Comparison: Molnupiravir vs Placebo; Adjusted differences and the corresponding confidence intervals are based on Miettinen & Nurminen method stratified by age and household size; Test type: Superiority; p = 0.0848, Miettinen & Nurminen method; Confidence Interval = -2, 95% CI 2-sided [-5 to 0.9]

2. Primary Outcome: Percentage of Participants With ≥1 Adverse Event
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: 29 days
Population: Safety Analyses was conducted in the APaT population, which consists of all randomized participants who received at least 1 dose of study intervention. Index participants were not included in OM analysis per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir | Placebo
Number analyzed (Participants) | 763 | 765
Participants | 94 | 105
Statistical Analysis 1: Comparison: Molnupiravir vs Placebo; 95% CIs (Tier 2 endpoints) was provided for between treatment differences in the percentage of participants with events; these analyses was performed using the Miettinen and Nurminen method; Test type: Other — Estimated differences and confidence intervals are provided; Miettinen & Nurminen method; Confidence Interval = -1.4, 95% CI 2-sided [-4.8 to 2.0]

3. Primary Outcome: Percentage of Participants Discontinuing From Study Therapy Due to AE
Description: as for outcome 2
Time Frame: Up to 5 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir | Placebo
Number analyzed (Participants) | 763 | 765
Participants | 3 | 1
Statistical Analysis 1: Comparison: Molnupiravir vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — Estimated differences and confidence intervals are provided; Miettinen & Nurminen method; Confidence Interval = 0.3, 95% CI 2-sided [-0.4 to 1.0]

4. Secondary Outcome: Percentage of Participants (Regardless of SARS-CoV-2 in Baseline NP Swabs) Who Developed COVID-19 (Laboratory-Confirmed SARS-CoV-2 Infection With Symptoms) Through Day 14
Description: Participants who experienced targeted symptoms of COVID-19 (e.g., cough, sore throat) and had NP swabs tested for SARS-CoV-2 using reverse-transcription polymerase chain reaction (RT-PCR).Efficacy analysis was conducted on the mITT (modified intent to treat) population consisting of all randomized participants who received at least 1 dose of study intervention.
Time Frame: Up to Day 14
Population: Index participants were not included in OM analysis per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir | Placebo
Number analyzed (Participants) | 763 | 764
Participants | 78 | 103
Statistical Analysis 1: Comparison: Molnupiravir vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0205, Miettinen & Nurminen method; Confidence Interval = -3.2, 95% CI 2-sided [-6.3 to -0.1]

5. Secondary Outcome: Percentage of Participants Who Had Undetectable SARS-CoV-2 in Baseline NP Swabs and Developed COVID-19 (Laboratory-Confirmed SARS-CoV-2 Infection With Symptoms) Through Day 29
Description: Participants who experienced targeted symptoms of COVID-19 (e.g., cough, sore throat) and had NP swabs tested for SARS-CoV-2 using RT-PCR. The efficacy analysis population was the mITT (modified intent to treat) population consisting of all randomized participants who received at least 1 dose of study intervention.
Time Frame: Up to Day 29
Population: Index participants were not included in OM analysis per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir | Placebo
Number analyzed (Participants) | 630 | 634
Participants | 51 | 65
Statistical Analysis 1: Comparison: Molnupiravir vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Adjusted differences and the corresponding confidence intervals; Miettinen & Nurminen method; Confidence Interval = -2.2, 95% CI 2-sided [-5.4 to 1.0]

6. Secondary Outcome: Percentage of Participants Who Had Undetectable SARS-CoV-2 in Baseline NP Swabs and Developed Detectable SARS-CoV-2 in NP Swabs on or Before Day 14
Description: All participants had NP swabs collected at screening and through Day 14 to test for SARS-CoV-2 using RT-PCR. Efficacy analysis was conducted on the mITT (modified intent to treat) population consisting of all randomized participants who received at least 1 dose of study intervention.
Time Frame: Up to Day 14
Population: Index participants were not included in OM analysis per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir | Placebo
Number analyzed (Participants) | 572 | 589
Participants | 65 | 85
Statistical Analysis 1: Comparison: Molnupiravir vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Adjusted differences and the corresponding confidence intervals; Confidence Interval = -3, 95% CI 2-sided [-6.9 to 0.8]

7. Secondary Outcome: Percentage of Participants Who Had Detectable SARS-CoV-2 in Baseline NP Swabs and Developed COVID-19 (Laboratory-confirmed SARS-CoV-2 Infection With Symptoms) Through Day 14
Description: Participants who experienced targeted symptoms of COVID-19 (e.g., cough, sore throat) and had NP swabs tested for SARS-CoV-2 using RT-PCR. Efficacy analysis was conducted on the mITT (modified intent to treat) population consisting of all randomized participants who received at least 1 dose of study intervention.
Time Frame: Up to Day 14
Population: Index participants were not included in OM analysis per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Molnupiravir | Placebo
Number analyzed (Participants) | 114 | 114
Participants | 35 | 47
Statistical Analysis 1: Comparison: Molnupiravir vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — Adjusted differences and the corresponding confidence intervals; Miettinen & Nurminen method; Mean Difference (Final Values) = -10.5, 95% CI 2-sided [-22.7 to 2.0]

ADVERSE EVENTS:
Time Frame: Up to Day 29
Description: All cause mortality (ACM) was analyzed in all randomized participants.Safety Analyses was conducted in all-participants-as-treated (APaT) population, which consisted of all randomized participants who received at least 1 dose of study intervention. Per protocol all-cause mortality and AE information was not collected for index cases.
Groups:
- MK-4482: Participants were treated with molnupiravir 800 mg every 12 hours (Q12H) on Days 1 to 5.
Arm/Group | MK-4482 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/768 | 1/771
Serious Adverse Events (participants affected / at risk) | 3/763 | 2/765
Other Adverse Events (participants affected / at risk) | 0/763 | 0/765
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-4482 (N=763) | Placebo (N=765)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT04939428/Prot_SAP_000.pdf